CLINICAL TRIAL: NCT02687958
Title: Phase II Randomized Multicenter Study of Everolimus as Maintenance Therapy for Metastatic Neuroendocrine Carcinoma With Pulmonary or Gastroenteropancreatic Origin
Brief Title: Study of Everolimus as Maintenance Therapy for Metastatic NEC With Pulmonary or Gastroenteropancreatic Origin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC 02/2014
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Neuroendocrine Carcinoma
Keywords: GEP/ NEC
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Everolimus 10mg (every cycle) until PD (Experimental): Patients with stable disease, partial response or complete response after 4- 6 cycles of induction chemotherapy with Cisplatin or Carboplatin plus Etoposide or alternative first line chemotherapy according with local practice will receive maintenance therapy with Everolimus 10mg every cycle (28days) until PD or unacceptable toxicity.
  Interventions: Drug: Everolimus
- B Observational (No Intervention): Patients in this arm will meet observation criteria

INTERVENTIONS:
Drug: Everolimus — Maintenance therapy
  Other Names: Afinitor
  Arms: A Everolimus 10mg (every cycle) until PD

SUMMARY:
Cisplatin and Etoposide is the standard of care in NEC originating from the gastro-intestinal tract and lung, based on retrospective studies.

Nevertheless the prognosis of this group of patients is still poor with median survival of less than 20 months.

Everolimus is an mammilian target of rapamycin (mTOR) inhibitor that has been demonstrated to be active in patients with well and moderately differentiated primitive neuroectodermal tumor (pNET).

Recently, the Investigators demonstrated that the mammilian target of rapamycin (mTOR) pathway is overexpressed in NEC.

Based on the activity of Everolimus in the treatment of patients with well and moderately differentiated p-NET and on the evidence that even poorly differentiated forms express the pathway of m-TOR is conceivable that Everolimus could be active even in NEC.

DETAILED DESCRIPTION:
A platinum based chemotherapy (Cisplatin or Carboplatin) plus Etoposide is the standard of care in NEC originating from the gastro-intestinal tract and lung, based on retrospective studies. In these clinical studies and in clinical practice the median number of cycle administered is six due to dose depending toxicity of platinum and to the concept of maximum response.

The expression of mTOR pathways was evaluated in gastroenteropancreatic - Neuroendocrine tumor (GEP-NEC).

The Investigator found that 6/9 (67%) of poorly differentiated GEP-NEC evaluated expressed p mTOR. Interestingly this expression was not observed in small cell carcinoma (10).

Recently, was demonstrated that the mTOR pathway is overexpressed in NEC (11). Based on the activity of Everolimus in the treatment of patients with well and moderately differentiated p-NET and on the evidence that even poorly differentiated forms express the pathway of m-TOR is conceivable that Everolimus could be active even in NEC. In particular we want to test the hypothesis that a maintenance therapy (or an early second line) with Everolimus 10 mg/daily in non progressive patients after first line chemotherapy could improve outcome prolonging progression free survival (PFS).

The NORDIC NEC study recently published retrospectively analyzed 305 patients with metastatic GI NEC (or unknown primary predominantly with GI metastases).

In this large retrospective study patients with Ki-67 < 55% are less responsive to platinum based chemotherapy but have a longer survival than patients with Ki-67 > 55%; then Ki-67 < 55% is a positive prognostic factor and a negative predictive factor to platinum based chemotherapy (7).

These data indicate that GI-NEC might be not consider as a unique entity, even if they are all classified as G3 according to WHO 2010 classification.

In this randomized Phase 2 trial the investigator want to evaluate the activity of Everolimus 10 mg/daily as maintenance therapy in patients with NEC and Ki-67 < 55%.

In fact this subgroup of NEC patients could benefit mostly from a maintenance treatment with Everolimus 10 mg/daily since they are less chemo responder and they show better prognosis as G1-G2 NET.

There is not a standard second line therapy for NEC patients treated with platinum based doublet, nevertheless Temozolamide and Capecitabine (TX) represent a regimen used in this setting, based on small and retrospective series (8). Therefore in our study we recommend that all patients at first progression (even if out of the study) will receive TX (Capecitabine 750 mg/m2 po BID days 1-14 plus Temozolomide 200 mg/m2 po quaque die (QD) days 10-14 q28) in order to homogenize second line treatment. However, second line treatment is chosen by single investigators.

The aim of this study is to evaluate the activity of a maintenance therapy (or early second line) with Everolimus 10 mg daily in patients with stable disease, partial response or complete response after 6 cycles of induction chemotherapy with Cisplatin or Carboplatin plus Etoposide or alternative first line chemotherapy administered according to clinical practice.

The primary endpoint is progression free survival (PFS) defined as the time between randomization and the first evidence of progressive disease or date of death, whichever occurs first. Documentation of disease progression will be defined as per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria based on investigator assessment. The censoring date for a patient who is known to be progression-free would be the date of the last tumor assessment.

Secondary objectives are :

* Overall survival (OS) defined as the time from randomization to death from any cause
* Safety profile: Safety of the treatment will be evaluated by serious and non serious adverse events (AEs). AEs will be graded according to the Common Toxicity Criteria for Adverse Effects (CTCAE v4.03)
* Evaluation of prognostic/predictive factors on tumoral tissue of patients treated with maintenance everolimus 10 mg/daily. The expression of mTOR and kinases involved in its pathway will be assessed by immunohistochemistry (IHC)
* Detection and count of circulating tumor cells (CTCs) from peripheral blood samples by VERIDEX® and correlation between CTCs number and outcome of patients in terms of PFS and OS
* Detection of circulating tumor DNA (ctDNA) and correlation between ctDNA levels and and outcome of patients in terms of PFS and OS. Evaluation of mTOR pathway genes mutations on ctDNA

This study population will comprise subjects diagnosed with GEP-NEC or large-cells neuroendocrine carcinoma of the Lung with Ki67< 55% with stable disease, partial of complete response after 6 cycles of first line chemotherapy.

Adverse Event: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values (as specified by the criteria below), regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE. A diagnosis or syndrome should be recorded on the AE page of the case report form (CRF) rather than the individual signs or symptoms of the diagnosis or syndrome.

Disease progression is not to be reported as an AE. An overdose, accidental or intentional, whether or not it is associated with an AE, or abuse, withdrawal, sensitivity or toxicity to an investigational product should be reported as an AE. If an overdose is associated with an AE, the overdose and adverse event should be reported as separate terms.

All subjects will be monitored for AEs during the study. Assessments may include monitoring of any or all of the following parameters: the subject's clinical symptoms, laboratory, pathological, radiological or surgical findings, physical examination findings, or other appropriate tests and procedures.

All AEs will be recorded by the Investigator from the time the subject signs informed consent to at least 30 days after the last dose of CT or until the last study visit, whichever period is longer. Adverse Events and serious adverse events (SAEs) will be recorded on the AE page of the CRF and in the subject's source documents. All SAEs must be reported to PIs within 24 hours of the Investigator's knowledge of the event by facsimile, or other appropriate method, using the SAE Report Form, or approved equivalent form. All SAEs will be also reported to Novartis safety desk within 15 days of learning.

Serious adverse events will be summarized.

Safety analyses: All pats who receive at least 1 dose of study drug will be evaluated for safety and toxicity. Adverse event (AE) terms and severity grades will be assigned by the investigator using CTCAE v. 4.03.

Safety analyses will include listings and/or summaries of the following:

* Treatment emergent adverse events (TEAEs), including seriousness, severity and possible relationship to study drug
* Dose adjustments
* CTCAE grades for laboratory and non laboratory parameters

Number of Patients: Thirty pts (20 in experimental arm and 10 in the control arm) will be randomized

Statistical method: This is an open-label study. Patients who meet all inclusion/exclusion criteria for enrollment will be allowed to enroll in the study. Those patients entering the study during all the trial will be allocated to arm A or arm B. Assignment to treatment will be determined prior to Cycle 1 d1 using an interactive response system by mail at a central location. Patients will be sequentially allocated to arm A or arm B with a 1:2 ratio.

This is a phase II study not powered for statistical comparison between arm A and B. The number of patients is sufficient for an exploratory analysis of the activity of Everolimus as maintenance therapy in this setting of patients. Only if the results in this analysis will be encouraging, a second step of the study will be powered for a comparison between arm A and B.

ELIGIBILITY:
Inclusion Criteria:

* Histological / cytological diagnosis of GEP Neuroendocrine Carcinoma (NEC) with Ki67< 55% (WHO 2010)
* Histological/cytological diagnosis of large-cells neuroendocrine carcinoma of the lung with Ki67 <55%;
* Stable disease, partial response or complete response (Recist 1.1) after 6 cycles of first line chemotherapy with Cisplatin plus Etoposide or alternative first line chemotherapy according with local practice
* non functional NEC
* locally advanced inoperable or metastatic disease
* measurable or evaluable disease according to RECIST criteria (version 1.1)
* Age> 18;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Adequate bone marrow function (Hb> 9.0 g / dL, absolute neutrophil count> 1.5 x 109 / L, platelets> 100 x 109 / L), renal function (serum creatinine <2 mg / dL x upper limit of normal (ULN) or creatinine clearance, Cockroft formula, ≥ 30 ml / min), hepatic function (serum bilirubin <1.5 x ULN, serum transaminases <2.5 x ULN in the absence of liver metastases or <5x ULN in the presence of liver metastases);
* Negative pregnancy test or breastfeeding women during childbearing age;
* Written informed consent;
* Approval of the Ethics Committee that will be required.

Exclusion Criteria:

* clinically significant cardiovascular disorders in the 6 months prior to randomization (congestive heart failure, myocardial infarction, unstable angina, severe uncontrolled cardiac arrhythmia, arterial thrombosis, cerebrovascular accidents, pulmonary thromboembolism);
* Functional Neuroendocrine Carcinoma NEC
* Neuroendocrine carcinoma with ki 67 > 55%
* ongoing uncontrolled infection;
* Concomitant intake of:

  * Drugs incompatible with concomitant everolimus;
  * Any other drug in clinical trials;
* History of other malignancy except carcinoma in situ of the cervix or basal / squamous cell carcinoma of the skin adequately treated;
* Presence of brain metastases;
* Any other serious or uncontrolled concurrent disease conditions that the safe administration of medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  progression free survival (PFS)

SECONDARY OUTCOMES:
OS | 24 months
  Overall survival (OS)
ctDNA | 24 months
  circulating DNA

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Di Costanzo, MD, Principal Investigator — AOU Careggi; Lorenzo Antonuzzo, MD, Principal Investigator — AOU Careggi
Locations (5):
- Italy (5):
  - S.C. Oncologia - Policlinico, Modena, Emilia-Romagna
  - U.O. Oncologia Medica 1 - AOU Pisana, Pisa, Tuscany
  - Azienda Ospedaliera "Spedali Civili di Brescia", Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Europeo di Oncologia, Milan

IPD SHARING:
Plan to Share IPD: Undecided